CLINICAL TRIAL: NCT04102163
Title: A Multicentre Prospective Observational Study to Assess Health Related Quality of Life in Crohn's Disease Patients With Complex Perianal Fistula Before and After Treatment: the CALYPSO Study
Brief Title: Health-Related Quality of Life in Crohn's Disease Participants With Complex Perianal Fistula Before and After Treatment
Acronym: CALYPSO
Status: Terminated | Type: Observational
Why Stopped: Business Decision; No Safety or Efficacy Concerns
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IBD-5008; U1111-1232-1975 (Registry Identifier: WHO)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Crohn Disease; Inflammatory Bowel Disease; Gastrointestinal Diseases; Intestinal Diseases
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Gastrointestinal Diseases; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants diagnosed with CD and CPF from approximately 20 Spanish hospitals, who will initiate medical or surgical treatment for their CPF within the eligibility period from Sep 2020 to Sep 2021, will be observed prospectively for approximately 31 months.

SUMMARY:
The purpose of this study is to assess the impact of treatment (medical and/or surgical) on Health-related Quality of Life (HRQoL) in participants with Crohn's Disease (CD) and Complex Perianal Fistula (CPF), by the Quality of Life in patients with Anal Fistula Questionnaire (QoLAF-Q), at 12 months after treatment initiation in routine clinical practice.

DETAILED DESCRIPTION:
This is a prospective follow-up post-authorization observational study of participants with CD and CPF. The study will provide real-world data on how CPF treatments in CD participants affect their HRQoL.

The study will enroll approximately 300 participants. All participants will be enrolled in one observational cohort.

This multi-center trial will be conducted in Spain. The study will collect data from a routine medical practice visits for CD participants with CPF and an application that will be designed ad hoc and will passively record participant's data. The overall duration of this study will be approximately 31 months. Participants will be followed up at Months 6 and 12 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with CD and CPF (defined as a fistula meeting any of the following criteria: high location [high intersphincteric, high transsphincteric, extrasphincteric, or suprasphincteric], multiple external openings, perianal abscess, anal stenosis, or proctitis).
2. Has tried and failed at least one prior treatment for CPF.
3. Starting a new pharmacological or surgical treatment for CPF.

Exclusion Criteria:

1. Diagnosed with indeterminate/unspecified type of inflammatory bowel disease (IBD).
2. Diagnosed with ulcerative colitis.
3. Diagnosed with fistula other than CPF (example rectovaginal).
4. Treated with darvadstrocel or other stem cells-based therapies within the eligibility period.
5. Previous fecal incontinence.
6. Lost to site follow-up for reasons other than death.
7. Participates or plans to participate in any interventional clinical trial.
8. Non fluent in Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with CD and CPF, who will initiate medical or surgical treatment for their CPF within Sep 2020 to Sep 2021, will be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Change From Baseline in QoLAF-Q Scores at Month 12 After Treatment Initiation for CPF | Baseline and Month 12
  QoLAF-Q evaluates quality of life (QoL) among participants with both simple and complex anal fistula (AF). It is composed of a total of 14 items with a Likert scale from 1 to 5 points. Its score range is the following: zero impact=14 points; limited impact=15 to 28 points; moderate impact=29 to 42 points; high impact=43 to 56 points; and very high impact=57 to 70 points.

SECONDARY OUTCOMES:
Number of Participants With Change From Baseline in QoLAF-Q Scores at Month 6 After Treatment Initiation for CPF | Baseline and Month 6
  QoLAF-Q evaluates QoL among participants with both simple and complex AF. It is composed of a total of 14 items with a Likert scale from 1 to 5 points. Its score range is the following: zero impact=14 points; limited impact=15 to 28 points; moderate impact=29 to 42 points; high impact=43 to 56 points; and very high impact=57 to 70 points.
Percentage of Participants With Clinically Significant Change From Baseline in QoLAF-Q Score at Months 6 and 12 After Treatment for CPF | Baseline, Months 6 and 12
  QoLAF-Q evaluates QoL among participants with both simple and complex AF. It is composed of a total of 14 items with a Likert scale from 1 to 5 points. Its score range is the following: zero impact=14 points; limited impact=15 to 28 points; moderate impact=29 to 42 points; high impact=43 to 56 points; and very high impact=57 to 70 points.
Change From Baseline in EuroQoL-Five Dimensions, Five Levels (EQ-5D-5L) Scores at Months 6 and 12 After Treatment for CPF | Baseline, Months 6 and 12
  The EQ-5D- is a generic, self-reported measure of utility that consists of a five-item descriptive system and a visual analogue scale (EQ VAS). The descriptive system has two versions, namely the 3L and 5L, both involving five health dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). In the EQ-5D-5L that will be used, participants may choose from the following five response levels: no problems=1; slight problems=2; moderate problems=3; severe problems=4; and unable to/extreme problems=5. Higher values indicate worst health.
Change From Baseline in Faecal Incontinence Quality of Life Scale (FIQOL) Scores at Months 6 and 12 After Treatment for CPF | Baseline, Months 6 and 12
  FIQOL comprises of 29 items that cover four dimensions of perceived health: lifestyle (10 items), behavior (9 items), depression/ self-perception (7 items), and embarrassment (3 items). Each item has a range of 1 to 4, with 1 being the lowest value for the state of quality of life.
Change From Baseline in Perceived Stress Scale (PSS) Scores at Months 6 and 12 After Treatment for CPF | Baseline, Months 6 and 12
  The PSS assesses participant's perceived nonspecific stress in a given situation or a daily life situation. The overall score of the scale is measured on a 14-item scale (from 0 to 4 points). Each item is scored 0 (never) to 4 (very often). Total score is obtained by inverting the scores on items 4, 5, 6, 7, 9, 10 y 13 (as follows: 0=4, 1=3, 2=2, 3=1 y 4=0) and summing up the scores of the 14 items. Higher total scores indicate higher perceived stress.
Change From Baseline in International Index of Erectile Function (IIEF) Scores at Months 6 and 12 After Treatment for CPF | Baseline, Months 6 and 12
  The IIEF is a multi-dimensional, self-administered questionnaire to assess erectile dysfunction. A score of 0 to 5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: Erectile Function (EF), Orgasmic Function (OF), Sexual Desire (SD) and Intercourse Satisfaction (IS). EF has five categories: 1-10(Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction). OF: sum of Questions (Q) 9 and Q10, each rated 0 (no sexual stimulation) to 5 (almost always/always). OF domain score range: 0 to 10; lower scores denoted lower OF. SD: sum of Q11 and Q12, each rated 1 (almost never or low/no sexual desire) to 5 (almost always or very high sexual desire). SD domain score range: 2 to 10;lower scores denoted lower SD. IS: sum of Q6, Q7, and Q8, each rated 0 (low/no satisfaction) to 5 (high satisfaction). IS domain score range: 0 to 15; lower scores denoted lower satisfaction.
Change From Baseline in Female Sexual Function Index (FSFI) Scores at Months 6 and 12 After Treatment for CPF | Baseline, Months 6 and 12
  The FSFI is a 19-item multidimensional self-report questionnaire for the assessment of female sexual function. It has five domains of sexual function, including: desire and subjective arousal, lubrication, orgasm, satisfaction, and pain/discomfort. FSFI is scored on a scale ranging from 1.2 to 6.0 (desire), 0 to 6.0 (arousal, lubrication, orgasm, and pain/discomfort) or 0.8 to 6.0 (satisfaction), with higher scores indicating better performance. The total score, falling in a possible range from 2.0 to 36.0, is obtained by adding the six domain scores together.
Number of Participants Based on Type of Treatment, Dose, Dose Frequency and Date of Initiation | Baseline
Number of Participants Based on Biological Data | Baseline, Months 6 and 12
  Biological data includes blood count, electrolytes, C-reactive protein (CRP), and fecal calprotectin.
Number of Participants With Comorbidities Based on Charlson Comorbidity Index | Baseline
  The Charlson Comorbidity Index is a 19-item measure assessing comorbid conditions. The total possible score on the Charlson Comorbidity Index ranges from 0 to 37. If a condition is not present, the score for that condition is zero. The higher scores indicate greater comorbidity.
Number of Participants With Comedications for Treatment of CD and Fistula | Baseline
Number of Participants With Target CPF | Baseline
Number of Participants With the Presence of new CPF at Months 6 and 12 | Months 6 and 12
Montreal Classification Assessed at Baseline | Baseline
  Montreal Classification includes age at diagnosis, disease location and disease behavior. Disease behavior was classified according to the following: B1 = non-stricturing, non-penetrating; B2 = structuring; B3 = penetrating; P = perianal disease modifier. The change in Montreal Classification is presented in three categories: no change, deterioration, and improvement. Deterioration defined as an increase in behavior index between 1 and 3, or development of perianal disease.
Number of Participants With Clinical characteristics Based on Harvey Bradshaw Index (HBI) | Baseline, Months 6 and 12
  HBI score is used to measure the disease activity of CD. It consists of clinical parameters: general well-being (0-4, where higher score means lower well being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools, where higher scores indicating more severe disease.
Number of Participants With Clinical Characteristics Based on Perianal Crohn´s Disease Activity Index (PDAI) or Fistula Drainage Assessment (FDA) | Baseline, Months 6 and 12
  The PDAI is a scoring system to evaluate the severity of perianal lesion associated with CD. It includes the following 5 items: (a) Discharge; (b) Pain; (c) Restriction of sexual activity; (d) Type of perianal disease; and (e) Degree of induration. Each item is graded on a 5-point scale ranging from no symptoms (score of 0) to severe symptoms (score of 4) and total range of score is from 0 to 20. Higher score means more severe disease.
Number of Occurrences of Treatment Switching or Dose Change | Months 6 and 12
Relation Between Participants QoLAF-Q Score and Clinical Variables | Baseline
  A parametric test will be used to measure the degree of association between the QolAF score and clinical variable. QoLAF-Q evaluates QoL among participants with both simple and complex AF. It is composed of a total of 14 items with a Likert scale from 1 to 5 points. Its score range is the following: zero impact=14 points; limited impact=15 to 28 points; moderate impact=29 to 42 points; high impact=43 to 56 points; and very high impact=57 to 70 points.
Number of Participants Based on Methods Used to Evaluate the Response to Different Treatments for CPF in Routine Clinical Practice | Months 6 and 12
Number of Participants Based on Effectiveness of Different Treatment Options for CPF Grouped According to Therapeutic Class | Months 6 and 12
  The effectiveness of different treatment options for CPF grouped according to therapeutic class (medical treatment, surgery or both) will be defined as the absence of draining despite gentle finger compression.
Health Care Resources Utilization (HCRU) | Baseline, Months 6 and 12
  HCRU includes emergency department and Intensive Care Units (ICU) visits; hospitalization (greater than or equal to (>=) 24 hours or related complications; number, type and reason for gastroenterology specialist or other specialty referral outpatient visits for management of complex perianal fistulas; surgeries or related complications; number of Magnetic Resonance Imaging (MRI) of the pelvis or transperineal, endoscopic ultrasound (EUS), and other non-surgical procedures performed to guide therapy, number of blood tests performed.
Correlation Between the Change in CD Participant's Scores in the QoLAF-Q, the EQ-5D-5L and Rapid Assessment Faecal Incontinence Score (RAFIS) | Baseline, Months 6 and 12
  Correlations between the scores obtained in the QoLAF-Q scale and the scores obtained in the RAFIS and EQ-5D-5L will be studied using Pearson correlation coefficients. QoLAF-Q evaluates QoL among participants with both simple and complex AF. It consists of a total of 14 items with a Likert scale from 1-5 points. Its score ranges:zero impact=14 points;limited impact=15 to 28 points; moderate impact=29 to 42 points;high impact=43 to 56 points;and very high impact=57 to 70 points. The EQ-5D- is a generic, self-reported measure of utility that consists of a 5-item descriptive system and EQ VAS. The descriptive system has 2 versions: 3L and 5L,both involving 5 health dimensions (mobility,self-care,usual activities, pain/discomfort and anxiety/depression). In the EQ-5D-5L that will be used, participants may choose from the following 5 response levels:no problems=1; slight problems=2;moderate problems=3; severe problems=4;and unable to/extreme problems=5.Higher values indicate worst health.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (20):
- Spain (20):
  - Hospital Reina Sofia, Córdoba, Andalusia
  - Hospital San Cecilio, Granada, Andalusia
  - Hospital Universiario Juan Ramon Jimenez, Huelva, Andalusia
  - Hospital Regional de Malaga, Málaga, Andalusia
  - Hospital Virgen del Rocio, Seville, Andalusia
  - Hospital Nuestra Senora de la Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Universitario Rio Hortega, Valladolid, Castille and León
  - Hospital Santa creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Vall d'Hebron, Barcelona, Catalonia
  - Hospital Parc Tauli, Barcelona, Catalonia
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Complejo Hospitalario Universitario de Ferrol, A Coruña, Galicia
  - Complejo Hospitalario de Pontevedra, Pontevedra, Galicia
  - Hospital de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Gregorio Maranon, Madrid, Madrid
  - Fundacion Jimenez Diaz, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/